CLINICAL TRIAL: NCT00951080
Title: Lower Extremity Venous and Diabetic Ulcer Negative Pressure Wound Therapy Trial.
Brief Title: SNaP Wound Care System Versus Traditional NPWT Device for Treatment of Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNP041609
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Ulcers; Wounds
Keywords: ulcer; venous; diabetic; wounds and injuries
MeSH Terms: conditions — Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SNaP Wound Care System (Experimental)
  Interventions: Device: SNaP Wound Care System
- Traditional NPWT System (Active Comparator)
  Interventions: Device: Traditional NPWT System

INTERVENTIONS:
Device: Traditional NPWT System — Standard wound dressing applications followed by negative pressure system application per manufacturer recommendations.
  Arms: Traditional NPWT System
Device: SNaP Wound Care System — Wound dressing applications using customized system. Dressing applications changes per manufacturer recommendation.
  Arms: SNaP Wound Care System

SUMMARY:
The purpose of this study is to evaluate a novel negative pressure wound therapy (NPWT) device called the SNaP device compared to a traditional NPWT device for the treatment of lower extremity diabetic and venous ulcer wounds.

DETAILED DESCRIPTION:
This is a prospective, randomized, two-arm, non-inferiority, multi-center study comparing negative pressure therapy wound healing outcomes between the SNaP Wound Care System and traditional NPWT systems.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Venous Ulcer or Diabetic Ulcer with a surface area < 100 sq. cm and < 10 cm in widest diameter on lower extremity, but larger than 1 sq. cm
* Subject has wound present for >30 days despite appropriate wound care
* Subject has adequate blood perfusion (Defined as either transcutaneous oxygen measurements of the dorsum of the foot >30 mmHg or 0.7 < ABI <1.2)
* Subject has wound in location amendable to creation of airtight seal around wound using NPWT dressings
* Subject is able to understand and provide written consent
* Subject able to understand and provide written consent
* Male or non-pregnant female willing to have urine pregnancy test

Exclusion Criteria:

* Subject has Active Infection (Redness, Swelling, Pain, Purulent Exudate)
* Subject has Untreated Osteomyelitis
* Subject has Allergy to Wound Care Products used in the study
* Subject has Malignancy, Burn, Collagen Vascular Disease, Sickle Cell, Vasculopathy, or Pyoderma Gangrenosum Origin of Wound
* Subject has Active Charcot Arthropathy of the Foot
* Subject has study wound location on toes or plantar surface of foot
* Subject has uncontrolled hyperglycemia (HbA1C >12%)
* Subject has end stage renal disease requiring dialysis
* Subject is undergoing active chemotherapy treatment that inhibits wound healing
* Subject has had previous treatment with NPWT device, growth factors, hyperbaric oxygen, or bioengineered tissue product within 30 days of enrollment
* Subject has a >30% wound surface area reduction in size at 1 week after screening visit
* Subject has any other condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study
* Subject is unwilling or unable to comply with protocol requirements
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM, Ph.D., Principal Investigator — Southern Arizona Limb Salvage Alliance (SALSA)
Locations (17):
- United States (17):
  - Hope Research Institute, Phoenix, Arizona
  - Southern Arizona Limb Salvage Alliance (SALSA), Tucson, Arizona
  - Center for Clinical Research, Inc., Castro Valley, California
  - Jay Mukker, DPM Inc., Fresno, California
  - Palomar Pomerado Health Wound Care Center, Poway, California
  - O'Connor Wound Care Clinic, San Jose, California
  - John Muir Wound Care Center, Walnut Creek, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Bethesda Health City Wound Care Center, Boynton Beach, Florida
  - Wound Care on Wheels, LLC, Jacksonville, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Weil Foot & Ankle Institute, Des Plaines, Illinois
  - LA Cardiovascular & Limb Salvage Center, Lafayette, Louisiana
  - University of North Carolina, Chapel Hill, North Carolina
  - The Christ Hospital, Wound Healing Center, Cincinnati, Ohio
  - New Bridge Medical Research Corporation, Warren, Pennsylvania
  - Southwest Washington Medical Center Wound Healing Center, Vancouver, Washington

REFERENCES:
- [Result] Armstrong DG, Marston WA, Reyzelman AM, Kirsner RS. Comparison of negative pressure wound therapy with an ultraportable mechanically powered device vs. traditional electrically powered device for the treatment of chronic lower extremity ulcers: a multicenter randomized-controlled trial. Wound Repair Regen. 2011 Mar-Apr;19(2):173-80. doi: 10.1111/j.1524-475X.2010.00658.x. PMID 21362084

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNaP Wound Care System | Traditional NPWT System
Started | 64 | 68
Completed | 38 | 41
Not Completed | 26 | 27
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Other | 19 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SNaP Wound Care System | Traditional NPWT System | Total
Number analyzed (Participants) | 64 | 68 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (14.2) | 65.6 (15.6) | 65.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 58
  Male | 31 | 43 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity (White) | 44 | 43 | 87
  Unknown | 20 | 25 | 45
Region of Enrollment [Number; unit: participants]
  United States | 64 | 68 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Wound Area
Description: The percent change in wound area as measured from Visitrak tracings (Value at 16 weeks minus value at baseline / value at baseline)
Time Frame: Baseline and 16 weeks
Measure: Median (Full Range); unit: percentage of baseline wound area
Arm/Group | SNaP Wound Care System | Traditional NPWT System
Number analyzed (Participants) | 59 | 56
percentage of baseline wound area | -85.7 [-100 to 392.3] | -94 [-100 to 500]

ADVERSE EVENTS:
Arm/Group | SNaP Wound Care System | Traditional NPWT System
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/64 | 2/68
Other Adverse Events (participants affected / at risk) | 14/64 | 18/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SNaP Wound Care System (N=64) | Traditional NPWT System (N=68)
Infection of study wound (Venous Leg Ulcer) (Infections and infestations) | 0 | 1
Cellulitis right foot (Venous Leg Ulcer) (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SNaP Wound Care System (N=64) | Traditional NPWT System (N=68)
Maceration (Skin and subcutaneous tissue disorders) | 10 | 13
Allergic reaction to dressing (Skin and subcutaneous tissue disorders) | 4 | 5
Pain (wound) (General disorders) | 1 | 4
Blisters (Skin and subcutaneous tissue disorders) | 3 | 4
Infection (Infections and infestations) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No